CLINICAL TRIAL: NCT06319053
Title: The Turbine-based Insufflator: a Safety and Feasibility Study During Laparoscopy.
Brief Title: The Turbine-based Insufflator Safety and Feasibility Study
Acronym: TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Politecnico di Milano University (Unknown); Health∼Holland, Topsector Life Sciences & Health (Unknown); Spatium Medical B.V. (Unknown); IDE Group B.V. (Unknown)
Responsible Party: Principal Investigator, Ass. Prof. J (John) Vlot MD, PhD, FEBPS, Consultant pediatric surgeon, Erasmus Medical Center
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: NL85402.078.23
Record Dates: First submitted 2024-02-15; First posted 2024-03-19 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Laparoscopy; Pneumoperitoneum
Keywords: Pneumoperitoneum; Device development; Insufflator; Laparoscopy
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Intervention Model Description: Consecutive patients from who informed consent can be acquired. The number of twelve participants was determined in conjunction with the Ethical Board of Erasmus MC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopy (Experimental): Adult study participants who are planned to undergo intraperitoneal laparoscopic surgery
  Interventions: Device: Turbine-based insufflator

INTERVENTIONS:
Device: Turbine-based insufflator — The use of a turbine-based insufflator instead of a conventional insufflator

SUMMARY:
The turbine-based insufflator for minimal access surgery provides a new technological basis for minimal invasive surgery insufflation. Turbine technology permits highly accurate pressure control, an intra-abdominal volume that is dynamically adapted to ventilation, and oscillometric measurements of abdominal compliance. This first-in-human study aims to evaluate technologic feasibility in terms of pressure stability performance and the safety of the device.

DETAILED DESCRIPTION:
The turbine-based insufflator for minimal access surgery provides a new technological basis for insufflation. Until now, insufflation uses a static pressurized gas volume that is strongly affected by external pressure and vice versa pressures onto the surrounding structures. Turbine technology permits highly accurate pressure control, and an intra-abdominal volume that is dynamically adapted to ventilation. In this safety and feasibility trial, the pressure stability of a turbine-based insufflator is investigated in patients undergoing laparoscopic surgery. In addition, small amplitude oscillation are superimposed to the intra-abdominal pressure at the start of insufflation. Those oscillometric measurements will be used to estimate the abdominal compliance through the forced oscillation technique.

Study population: Adults who are scheduled for an elective intraperitoneal laparoscopic surgical procedure at Erasmus MC.

Main study parameters: safety and feasibility of turbine-based insufflation in terms of (Serious) Adverse Device Effects.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Elective laparoscopic surgery
* Intraperitoneal procedure
* Planned use of a main 11 mm trocar
* Informed consent

Exclusion Criteria:

* Pregnancy
* Inability to contain the insufflation gas to the intraperitoneal cavity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of (serious) adverse device effects [Safety and feasibility of the device] | During the surgical procedure
  Recording all adverse device effects as defined in the study protocol

SECONDARY OUTCOMES:
Observation of insufflation pressure stability by continuously monitoring and recording. | During the surgical procedure
  Assessment of stability of the intra-abdominal pressure generated by the device during the surgical procedure using descriptive statistics of deviation from set-pressure.
Gas volume exchange | During the surgical procedure
  Determination of the gas volume exchange required to keep insufflation pressures stable.
Estimation of the abdominal compliance | <6 months after the surgical procedure
  During the surgical procedure, oscillometry is performed with different frequencies and different pressures. Based on the acquired data the abdominal cavity's compliance will be determined by calculating the Impedance.
Intra-abdominal target pressure in relation to the abdominal compliance | <6 months after the surgical procedure
  The target intra-abdominal pressure for the procedure as determined by the surgeon will be plotted on the compliance curve that is measured with oscillometry. Ultimately we aim to determine biomechanical optimum pressure based on oscillometry data.

CONTACTS AND LOCATIONS:
Overall Officials: J. Vlot, MD, PhD, Principal Investigator — Erasmus MC, University Medical Center Rotterdam
Locations (1):
- Erasmus MC, University Medical Center Rotterdam, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No